CLINICAL TRIAL: NCT06638775
Title: RESEARCH PROJECT on the APPLICATION of FUNCTIONAL ELECTROSTIMULATION on the UPPER LIMB in MULTIPLE SCLEROSIS
Brief Title: Functional Electrostimulation on the Upper Lip in Multiple Sclerosis
Acronym: EM/2024
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COPTOCYL/2025; IO/102025 (Other: Universidad de Burgos)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Electrode Site Reaction; Therapy; Directly Observed Therapy
Keywords: fesia grasp; multiple sclerosis; multicampe; therapy
MeSH Terms: conditions — Directly Observed Therapy; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): The Fesia Grasp device is based on the superficial electrical stimulation of the forearm musculature to provoke flexion and extension movements of the wrist, thumb, index finger and fingers 3, 4 and 5.
  Interventions: Other: Fesia Grasp
- CONTROL GROUP (Experimental): Globus elite intervention: is an electro-stimulator designed for sport and fitness, but with special attention also for beauty treatments thanks to the new sequential stimulation currents, excellent for their draining effects.
  Interventions: Other: GLOBUS ELITE

INTERVENTIONS:
Other: Fesia Grasp — The Fesia Grasp device is based on the superficial electrical stimulation of the forearm musculature to provoke flexion and extension movements of the wrist, thumb, index finger and fingers 3, 4 and 5.
  Arms: EXPERIMENTAL GROUP
Other: GLOBUS ELITE — is an electro-stimulator designed for sport and fitness, but with special attention also for beauty treatments thanks to the new sequential stimulation currents, excellent for their draining effects.
  Arms: CONTROL GROUP

SUMMARY:
Multiple sclerosis (MS) is an autoimmune disease where immune cells attack the body, triggering an inflammatory response. A study comparing multifield FES and conventional FES on upper extremity motor skills and functional independence in MS patients will be conducted. Results suggest that both types of FES treatments normalize muscle tone, showing superior results compared to those without FES therapy. The study aims to compare the effects of both types on MS patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune disease in which cells of the immune system attack the body itself. This condition generates an activation of the immune system that triggers an inflammatory response. General objective: To compare the effect of multifield FES and conventional FES on upper extremity motor skills and functional independence in people with MS. Methodology: A three-arm prospective longitudinal multicenter randomized controlled trial (RCT) will be conducted: conventional therapy (Control Group, CG), an experimental group 1 (EG1) which in addition to this same treatment will use the conventional FES tool, through the Globus Elite device, and an experimental group 2 (EG2) which will differ from GE1 in that it will use the FES multi-field device through FESIA Grasp. Results: It is expected that people who have used any type of FES will have a more normalized muscle tone compared to those who have not received this type of treatment. The research compares the effects of two types of FES in people with multiple sclerosis, focusing on improved motor skills and functional independence. Both FES treatments are expected to normalize muscle tone, showing superior results compared to those who do not receive this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age and sign the informed consent form.
* Not suffer from any pathology in the upper limb such as tendinitis, oedema, fractures, etc.
* Intact skin (no breaks, scratches, cuts, and other superficial or deep injuries) on the arm where the devices will be placed if applicable

Exclusion Criteria:

* Severe medical problems.
* Use of a pacemaker.
* Pregnancy.
* Cutaneous neuropathies.
* Presence of other neuromuscular pathologies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Nine Hole Peg Test | 3 weeks
  The Nine Hole Peg Test (NHPT) (Mathiowetz et al, 1985), consists of a manual test, in which the subject must place 9 pegs in their corresponding 9 holes, and remove them again, the variable measured being the time it takes to carry out the whole process.
Box and Block | 3 weeks
  The Box and Block scale is a tool with standardised dimensions and materials. It specifies that the subject should sit in front of a rectangular box with his or her hands next to it. The box is constructed of wood with a base 53.7 cm wide and 25.4 cm long; it is divided into two square compartments of 25.4 cm each side separated by a 15.2 cm high divider; both compartments are padded in order to reduce noise during testing. The test contains 150 cube-shaped wooden blocks of 2.5 cm on each side. The number of blocks the subject has carried from one compartment to the other with each hand in one minute of time is to be recorded. Higher scores indicate better manipulative skills.
Jamar hand-held dynamometer | 3 weeks
  The Jamar hand dynamometer is used to measure grip strength in the hand, allowing the force exerted by the individual to be converted into a numerical reading. The subject is asked to grip the device and is instructed to perform the maximum sustained contraction. The force is recorded in kilograms.
Movement imagery Questionnaire, revisado (MIQ-RS) | 3 weeks
  The MIQ-RS questionnaire (Gregg et al, 2010) consists of 2 subscales, one visual and one kinaesthetic, of 7 items each, each item being scored on a 7-point Likert scale (the higher the score, the easier it is to imagine). For all items, the user is asked to perform a certain motor act (only once), to return to the starting position, and then to imagine it. When scoring the visual scale, the participant is asked to generate an image "as if they could see themselves" doing the gesture, while the kinaesthetic scale asks them to "recall the sensation of the movement".
Chronometry | 3 weeks
  Chronometry is defined as the temporal congruence between an executed motor act and the same imagined act.
  In this case, the NHPT itself is proposed as the motor act executed. So, once administered to obtain the test variable (time taken to perform), the participant will be asked to imagine the performance of the test, and both measures will be timed.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Hilario Ortiz phd, Principal Investigator — University of Burgos

IPD SHARING:
Plan to Share IPD: Yes
All participants will receive an informed consent form explaining the study to be carried out and the data to be used.
Supporting Information: ICF
Time Frame: Data will be available throughout the intervention with participants for 3 months.
Access Criteria: Being a study participant: each participant will be provided with a password to access their informed consent and the research protocol.

REFERENCES:
- [Background] Vázquez Sánchez F. Manual de neurología para terapia ocupacional. García López Beatriz, editor. Madrid: Editorial Medica Panamericana; 2023.